CLINICAL TRIAL: NCT04556149
Title: SARS-CoV-2/COVID-19 Study of the Audible and Inaudible Vibroacoustic E-stethoscope - imPulse™ Una
Brief Title: imPulse™ Una Full-spectrum, Over Clothing E-stethoscope
Status: Completed | Type: Observational
Sponsor: Level 42 AI, Inc. (Industry)
Collaborators: Schmidt Futures (Unknown); Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: 00110011
Record Dates: First submitted 2020-05-23; First posted 2020-09-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Corona Virus Infection; Coronavirus
Keywords: infrasound; e-stethoscope; biosignature; SARS-CoV-2/COVID-19
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Inpatients with confirmed COVID-19 with pulmonary symptoms
  Interventions: Device: imPulse™ Una e-stethoscope; Device: Philips Lumify Ultrasound System
- Matched Control: Inpatients without COVID-19 with non-pulmonary diagnoses or symptoms
  Interventions: Device: imPulse™ Una e-stethoscope; Device: Philips Lumify Ultrasound System

INTERVENTIONS:
Device: imPulse™ Una e-stethoscope — The imPulse™ System is an every/anywhere-point-of-care cardiopulmonary functional state assessment platform designed to capture normal and abnormal, audible and inaudible cardiopulmonary sounds, rhythms and patterns, via a real-time, intelligent, full-spectrum phonocardiogram obtained from direct to skin coupling or through a layer of clothing.
Device: Philips Lumify Ultrasound System — Point-of-care ultrasound

SUMMARY:
This study generates robust clinical data to train ML/AI algorithms of the Sponsor's imPulse™ Una full-spectrum e-stethoscope for digital diagnostic feature synthesis of symptomatic SARS-CoV-2/COVID-19 biosignatures for rapid and accurate mass screening.

DETAILED DESCRIPTION:
This study is designed to evaluate the ability of the imPulse™ Una e-stethoscope to differentiate vibroacoustic signals in inpatients with and without confirmed COVID-19 as the first step to establish the performance characteristics - sensitivity, specificity, positive and negative predictive value - of the imPulse™ Una device for early and rapid, point-of-care diagnosis of COVID-19. This will inform the utility and design of further larger-scale studies using the device.

ELIGIBILITY:
Inclusion Criteria

* Individuals hospitalized within a Johns Hopkins-affiliated hospital
* Able to understand and willingness to comply with study procedures
* Cases - inpatients with positive COVID-19 PCR test, collected from a respiratory sample within the last 7 days, AND pulmonary symptoms within 72 hours of enrollment
* Controls - inpatients without COVID-19 diagnosis and no pulmonary diagnosis or symptoms
* Cases or Control not able to sit or stand will be allowed to participate in just the parts of the staircase exam they're capable of doing.

Exclusion Criteria

* Assisted ventilation, including high flow nasal cannula, or ventilator support
* Unable to comply with study procedures, defined at investigator's discretion
* Participants with any visible skin infections or open wounds in areas where the imPulse™ Una device would be applied

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult men and women will be recruited from among hospitalized patients with symptomatic COVID-19 infection who are not receiving ventilator support. One hospitalized control without lung disease or pulmonary symptoms will be selected for each case.
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2020-12-02 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance characteristics | through study completion, an average of 2 weeks
  Sensitivity, specificity, positive and negative predictive values - of the imPulse™ Una device for point-of-care diagnosis of COVID-19.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Dooley, MD, PhD, Principal Investigator — Johns Hopkins School of Medicine; Ed Fuchs, MBA, Study Director — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dooley KE, Morimoto M, Kaszuba P, Krasne M, Liu G, Fuchs E, Rexelius P, Swan J, Krawiec K, Hammond K, Ray SC, Hafen R, Schuh A, Jumbe NLS. Evidence Generation for a Host-Response Biosignature of Respiratory Disease. Viruses. 2025 Jul 2;17(7):943. doi: 10.3390/v17070943. PMID 40733560